CLINICAL TRIAL: NCT01332786
Title: Phase 1 Study Evaluating the Tolerance and Biologic Activity of Intravenous Infusions of Tigecycline in Patients With Relapsed or Refractory AML
Brief Title: Safety Study Evaluating Intravenous Infusions of Tigecycline to Treat Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Kansas (Other); Memorial Sloan Kettering Cancer Center (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-029
Record Dates: First submitted 2011-03-31; First posted 2011-04-11 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tigecycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tigecycline (Experimental)
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — Dosage Form: one-hour intravenous infusion Dosage levels, frequency, duration: (3-week cycles)
  * Level 1: 50 mg daily x 10 doses; 1 week rest
  * Level 2: 100 mg daily x 10 doses; 1 week rest
  * Level 3: 150 mg daily x 10 doses; 1 week rest
  * Level 4: 200 mg daily x 10 doses 1 week rest
  * Level 5: 250 mg daily x 10 doses; 1 week rest
  * Level 6: 300 mg daily x 10 doses; 1 week rest
  * Level 7: 350 mg daily x 10 doses; 1 week rest
  Other Names: Tygacil

SUMMARY:
The purpose of this study is to determine whether tigecycline is safe and which dosage is most effective in the treatment of patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
Relapsed and refractory hematologic malignancies have poor responses to standard therapy and are associated with a poor prognosis. For example, relapsed acute myeloid leukemia (AML) is a highly aggressive and resistant disease, particularly when associated with first complete response (CR) duration of less than 12 months. Thus, there is an urgent need for new agents in relapsed and refractory hematologic malignancies such as acute leukemia. In elderly patients, where the tolerance of aggressive induction therapy is often poor and curative options such as bone marrow transplantation HSCT are not available, the need for effective non-aggressive drug regimens for AML is even greater.

Tigecycline is a glycylcycline derivative of tetracycline. Tigecycline is currently indicated for the treatment of complicated skin and skin structure infections, and complicated intra-abdominal infections. This clinical trial is a Phase I dose escalation study of tigecycline in patients with relapsed or refractory AML or those with newly diagnosed disease not eligible for induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of relapsed or refractory AML for which all potentially curative or standard salvage therapy options have been exhausted; OR AML without prior treatment who are not eligible for induction chemotherapy as defined as age > or equal to 80 or age > 70 with poor risk cytogenetics (3 or more abnormalities, -5/del(5q), 3q abnormalities, or -7) or stable co-morbidities that would preclude induction chemotherapy such as LVEF less than 40% and/or DlCO less than 60% expected
* ECOG 0-2 performance status
* Biochemical values within the following range
* Serum creatinine <2x upper limit of normal
* Total bilirubin <1.5x upper limit of normal
* AST and ALT <2x upper limit of normal
* Recovery from non-hematologic toxicity from prior chemotherapy
* Able and willing to provide informed consent

Exclusion Criteria:

* Allergy to tetracycline or minocycline
* Uncontrolled intercurrent illness such as uncontrolled diabetes or active uncontrolled infection
* Active systemic bacterial, fungal, or viral infection
* Concomitant use of linezolid or chloramphenicol that are known to inhibit mitochondrial protein synthesis
* Pregnant or breast feeding
* Known active CNS involvement with AML
* Neurologic symptoms related to uncontrolled illnesses or unexplained causes
* Psychiatric illness that would limit compliance with study
* Receiving systemic chemotherapy other than hydroxyurea to control circulating blast counts. Concomitant hydroxyurea is permitted, but only in the first cycle of therapy
* Prior therapy with tigecycline as an anti-cancer therapy or any use of the drug in the last month
* Use of other investigational anti-leukemic therapy within 14 days of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Toxicity evaluated according to CTCAE version 4.03 | Reviewed at each visit and assessed at the end of each 3-week cycle

SECONDARY OUTCOMES:
Response rate assessment of tigecycline through laboratory assessments | Assessed at the end of each 3-week cycle for the study duration
  Bone marrow assessment, absolute neutrophil count, platelet counts

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Schimmer, MD, Study Director — University Health Network, Toronto
Locations (3):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - The University of Kansas Medical Center, Kansas City, Kansas
- Princess Margaret Hospital, Toronto, Ontario, Canada